CLINICAL TRIAL: NCT05913830
Title: Effectiveness of Auricular Acupressure on the Methadone Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Ya-Fang Lin, National Taipei University of Nursing and Health Sciences, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TCHIRB-11012011
Record Dates: First submitted 2023-05-29; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Conditions:Effectiveness of Auricular Acupressure on the Methadone Patient

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: (Experimental): Experimental Group A total of 36 methadone patients will receive auricular pressure
  Interventions: Other: Auricular pressure
- Control group: (No Intervention): Control group 36 bits No interventions implemented

INTERVENTIONS:
Other: Auricular pressure — The seeds of blancia blanc were fixed on the acupoints with patches. The intervention measure in the experimental group was auricular point sticking. The two groups received four measurements before the intervention and 2 weeks, 4 weeks, and 6 weeks after the start; while the control group received no Auricular pressure.
  Arms: Experimental group:

SUMMARY:
This study aims to investigate the effect of auricular point sticking on constipation in patients with methadone

DETAILED DESCRIPTION:
This study is a randomized controlled trial, taking 72 methadone constipation patients from a hospital in the north as objects, and divided them into an auricular point group and a control group. The experimental group was given auricular point sticking, while the control group only used sticking cloth. The two groups were measured for constipation, TCM constitution, anxiety, depression and quality of life before the intervention and 2 weeks, 4 weeks, and 6 weeks after the start.

ELIGIBILITY:
Inclusion Criteria:

1. Methadone patients over 20 years old.
2. Those who have clear consciousness and can communicate in Chinese and Taiwanese.
3. The frequency of defecation is less than three times a week.
4. Willing to sign a written subject consent form.

Exclusions:

1. Those with wounds, broken skin, and blisters on the skin of both ears.
2. People with blood coagulation problems and related diseases, such as: purpura, hemophilia, etc.
3. Age <20 years old.
4. Subjects who use drugs to improve constipation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The effect of constipation after auricular acupressure | six weeks
  There were significant between-group differences in Bristol Stool Type at Weeks 2, 4, and 6 between the two groups (p= .003, p < .001, p < .001, respectively). The distribution of Bristol Stool Types in the second week, the fourth week, and the sixth week of the above-mentioned auricular point sticking intervention in the two groups all had statistically significant differences.
The effect of TCM constitution after the intervention of auricular acupressure | six weeks
  The total score of the experimental group in the 2nd week and the 6th week was damp and hot (p < .05); the experimental group had a significant difference in the decrease of the total score of the qi stagnation in the 4th week and the 6th week (p < .05).
The effect of intervention on depression and anxiety after auricular acupressure | six weeks
  There was no significant difference in the scores of the Bayesian Anxiety Scale and depression between the experimental group and the control group at the 2nd week, 4th week and 6th week (p > .05).
Effect of Interventional Auricular Acupressure on Quality of Life for Constipation | six weeks
  There were significant differences in the decrease of the total score of the experimental group in the 2nd week, 4th week and 6th week (p < .05, p < .001, p < .001 respectively)

CONTACTS AND LOCATIONS:
Locations (1):
- Ya-Fang Lin, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No